CLINICAL TRIAL: NCT04662255
Title: A Phase 3 Open-Label, Randomized Study of LOXO-305 Versus Investigator Choice of BTK Inhibitor in Patients With Previously Treated BTK Inhibitor Naïve Mantle Cell Lymphoma (BRUIN MCL-321)
Brief Title: Study of BTK Inhibitor LOXO-305 Versus Approved BTK Inhibitor Drugs in Patients With Mantle Cell Lymphoma (MCL)
Acronym: BRUIN-MCL-321
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Loxo Oncology, Inc. (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Organization: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18072; J2N-OX-JZNM (Other: Eli Lilly and Company); LOXO-BTK-20019 (Other: Eli Lilly and Company)
Expanded Access: NCT05172700 (Approved for marketing)
Record Dates: First submitted 2020-12-04; First posted 2020-12-10 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Lymphoma, Mantle-Cell
Keywords: Bruton's Tyrosine Kinase Inhibitor; BTKi; Hematologic Disease; Lymphoma, non-Hodgkin's; Lymphoma, B-Cell; Lymphoma; pirtobrutinib
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Hematologic Diseases; Lymphoma, Non-Hodgkin; Lymphoma, B-Cell; Lymphoma | interventions — pirtobrutinib; ibrutinib; acalabrutinib; zanubrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Pirtobrutinib) (Experimental): Orally
  Interventions: Drug: Pirtobrutinib
- Arm B (Ibrutinib, Acalabrutinib, or Zanubrutinib) (Active Comparator): Investigator's choice (based on local availability) of ibrutinib, acalabrutinib or zanubrutinib orally. Options are limited to those that are available/approved in the specific country.
  Interventions: Drug: Ibrutinib; Drug: Acalabrutinib; Drug: Zanubrutinib

INTERVENTIONS:
Drug: Pirtobrutinib — Oral
  Other Names: LOXO-305; LY3527727
  Arms: Arm A (Pirtobrutinib)
Drug: Ibrutinib — Oral
  Other Names: Imbruvica
  Arms: Arm B (Ibrutinib, Acalabrutinib, or Zanubrutinib)
Drug: Acalabrutinib — Oral
  Other Names: Calquence
  Arms: Arm B (Ibrutinib, Acalabrutinib, or Zanubrutinib)
Drug: Zanubrutinib — Oral
  Other Names: Brukinsa
  Arms: Arm B (Ibrutinib, Acalabrutinib, or Zanubrutinib)

SUMMARY:
This is a study for participants with a type of blood cancer called mantle cell lymphoma (MCL). The main purpose is to compare pirtobrutinib (LOXO-305) to other drugs that work in a similar way that have already been approved by the United States Food and Drug Administration (US FDA). Participation could last up to two years, and possibly longer, if the disease does not progress.

DETAILED DESCRIPTION:
This is a Phase 3 global, randomized, open-label study comparing pirtobrutinib (Arm A) to investigator's choice of ibrutinib, acalabrutinib or zanubrutinib (Arm B) in MCL patients who have received 1 or more lines of therapy and are BTK inhibitor naïve.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed MCL diagnosis
* Previously treated with at least one prior line of systemic therapy for MCL
* Measurable disease per Lugano criteria
* Eastern Cooperative Oncology Group (ECOG) 0-2
* Absolute neutrophil count ≥ 0.75 × 109/L without granulocyte-colony stimulating factor support within 7 days of screening
* Hemoglobin ≥ 8 g/dL not requiring transfusion support or growth factors within 7 days of screening
* Platelets ≥ 50 × 109/L not requiring transfusion support or growth factors within 7 days of screening.
* AST and ALT ≤ 3.0 x upper limit of normal (ULN)
* Total bilirubin ≤ 1.5 x ULN.
* Creatinine clearance of ≥ 30 mL/min according to Cockcroft/Gault Formula

Exclusion Criteria:

* Prior treatment with an approved or investigational BTK inhibitor
* History of bleeding diathesis
* History of stroke or intracranial hemorrhage within 6 months of randomization
* History of allogeneic or autologous stem cell transplant (SCT) or chimeric antigen receptor modified T-cell (CAR-T) therapy within 60 days of randomization
* Clinically significant cardiovascular disease
* Prolonged QT interval corrected using Fridericia's formula (QTcF) > 470 ms on 2/3 consecutive ECGs, and mean QTcF>470 ms on all 3 ECGs
* Known HIV infection or active HBV, HCV, or CMV infections. (Certain participants with controlled HBV infections may still be eligible)
* Clinically significant active malabsorption syndrome or other condition likely to affect gastrointestinal (GI) absorption
* Ongoing chronic treatment with strong cytochrome P450 3A4 (CYP3A4) inhibitors or inducers which cannot be stopped within 3-5 half lives of the CYP3A inhibitor therapy prior to start of study drug treatment.
* Patients requiring therapeutic anticoagulation with warfarin or another Vitamin K antagonist.
* Vaccination with live vaccine within 28 days prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2021-04-08 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
To compare progression-free survival (PFS) of pirtobrutinib as monotherapy (Arm A) to investigator choice of covalent BTK inhibitor monotherapy (Arm B) in patients with previously treated mantle cell lymphoma (MCL) | Up to approximately 24 months
  Assessed per Lugano criteria

SECONDARY OUTCOMES:
To compare Event Free Survival (EFS) as monotherapy (Arm A) to investigator choice of covalent BTK inhibitor monotherapy (Arm B) treatment arms | Up to approximately 24 months
  Defined as the time from randomization to progressive disease (PD) or start of new treatment for MCL or withdrawal from trial due to toxicity or death
To compare Time to Treatment Failure (TTTF) as monotherapy (Arm A) to investigator choice of covalent BTK inhibitor monotherapy (Arm B) treatment arms | Up to approximately 24 months
  Time from randomization to time when discontinuation criteria met
Time to worsening (TTW) of MCL-related symptoms | Up to approximately 24 months
  Using symptom questions identified from the European Organization for Research and Treatment of Cancer (EORTC) item library. The range of raw scores for these items could be from 0 to 52 with highest score being worse symptoms.
Comparative Tolerability as measured by proportion of time with high side effect burden | Up to approximately 24 months
  Using 18 items covering 10 Patient Reported Outcome- Common Terminology Criteria for Adverse Events (PRO-CTCAE) concepts for frequency (0-5 with 5 as most frequent), and/or presence (0-1 with 1 being present), or Severity (0-5 with 5 as most severe) and/or presence (0-1 with 1 being present); these selective adverse events will be framed and then overall side effect burden will be ascertained with the Functional Assessment of Cancer Therapy (FACT) - Item GP5. The range of this item is 0 -4 with 4 as most bothersome.
To compare Overall Response Rate (ORR) of pirtobrutinib as monotherapy (Arm A) to investigator choice of covalent BTK inhibitor monotherapy (Arm B) treatment arms | Up to approximately 24 months
  Assessed per Lugano criteria
To compare Duration of Response (DOR) of pirtobrutinib as monotherapy (Arm A) to investigator choice of covalent BTK inhibitor monotherapy (Arm B) treatment arms | Up to approximately 24 months
  Assessed per Lugano criteria
To compare Overall Survival of pirtobrutinib as monotherapy (Arm A) to investigator choice of covalent BTK inhibitor monotherapy (Arm B) treatment arms | Up to approximately 24 months
  Assessed by survival

CONTACTS AND LOCATIONS:
Overall Officials: Patient Advocacy, Study Director — Loxo Oncology, Inc.
Locations (189):
- United States (36):
  - Alaska Oncology and Hematology, LLC, Anchorage, Alaska
  - Arizona Oncology Associates, P.C. - HOPE, Phoenix, Arizona
  - UCLA Medical Center, Los Angeles, California
  - USO-Rocky Mountain Cancer Center, Denver, Colorado
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Oncology-Hematology Associates of West Broward, Tamarac, Florida
  - Florida Cancer Specialists East, West Palm Beach, Florida
  - University of Kentucky Markey Cancer Center, Lexington, Kentucky
  - Mercy Health-Paducah Medical Oncology and Hematology, Paducah, Kentucky
  - Tulane Cancer Center Office of Clinical Research, New Orleans, Louisiana
  - Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - DFCI Lymphoma, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University Medical School, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Messino Cancer Center, Asheville, North Carolina
  - Levine Cancer Institute, Charlotte, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Oncology Hematology Care Inc, Cincinnati, Ohio
  - Willamette Valley Cancer Institute & Research Ctr., Eugene, Oregon
  - Sarah Cannon Research Institute SCRI, Nashville, Tennessee
  - Texas Oncology-Austin Midtown, Austin, Texas
  - Texas Oncology - Bedford, Bedford, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Texas Oncology - McAllen, McAllen, Texas
  - Texas Oncology - Sherman, Sherman, Texas
  - US Oncology, The Woodlands, Texas
  - Texas Oncology - Tyler, Tyler, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - University of Virginia Health System, Charlottesville, Virginia
  - USO-Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
  - Froedtert Memorial Lutheran Hospital, Milwaukee, Wisconsin
- Australia (5):
  - The St. George Hospital, Kogarah, New South Wales
  - Royal Hobart Hospital, Hobart, Tasmania
  - Linear Clinical Research, Nedlands, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
  - Icon Cancer Care - The Wesley Medical Centre, Auchenflower
- Austria (2):
  - Uniklinikum Salzburg, Salzburg, Osterreich
  - Ordensklinikum Linz GmbH Elisabethinen, Linz, Upper Austria
- Belgium (3):
  - Universitair Ziekenhuis Gent, Ghent, Oost-Vlaanderen
  - AZ Delta, Roeselare, West Flanders
  - Universitaire Ziekenhuizen Leuven - Campus Gasthuisberg, Leuven
- Brazil (16):
  - Hospital São Lucas Copacabana, Rio de Janeiro, CEP
  - Hospital Beneficência Portuguesa de São Paulo, São Paulo, CEP
  - Centro de Oncologia e Hematologia do Ceará LTDA, Aldeota, Fortaliza
  - Hospital das Clínicas da UFGo - Goiânia, Goiânia, Goiás
  - Hospital Sao Domingos, São Luís, Maranhão
  - Instituto Nacional de Câncer - INCA, Rio de Janeiro, Rio de Jan
  - Centro de Pesquisa Clínica São Lucas, Campinas, Sau Paulo
  - Instituto de Ensino e Pesquisas São Lucas - IEP Hemomed, Pacaembu, São Paulo
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, Dept. CIP - Centro Integrado de Pesquisa, Rio Preto, São Paulo
  - CEPHO - Centro de Estudos e Pesquisas de Hematologia e Oncologia, Santo André, São Paulo
  - A. C. Camargo Cancer Center, São Paulo, São Paulo
  - HC - UFPR - Hospital de Clínicas da Universidade Federal do Paraná, Curitiba- PR
  - IPITEC, São Paulo
  - Hospital da Clinicas da Faculdade de Medicina da USP, São Paulo
  - Sociedade Beneficente Israelita Brasileira Hospital Albert Einstein, São Paulo
  - Hospital 9 De Julho, São Paulo
- Canada (3):
  - Cross Cancer Institute, Edmonton, Alberta
  - BC Cancer Vancouver, Vancouver, British Columbia
  - Cancer Care Manitoba, Winnipeg, Manitoba
- China (27):
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - Beijing ChaoYang Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Beijing Cancer hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Fujian Provincial Cancer Hospial, Fuzhou, Fujian
  - Cancer Center of Guangzhou Medical University, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Southern Medical University Nanfang Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Henan University of Science &Technology, Luoyang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Wuhan Union Hospital, Wuhan, Hubei
  - Yichang Central People's Hospital, Yichang, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Affiliated Tumor Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Lishui Central Hospital, Lishui, Zhejiang
  - Chongqing Cancer Hospital, Chongqing
  - Blood Institute of the Chinese Academy of Medical science, Tianjin
- Czechia (2):
  - Fakultni nemocnice Hradec Kralove, Hradec Králové, Hradec Králové
  - Fakultni nemocnice Brno, Brno
- Denmark (2):
  - Aarhus Universitetshospital, Aarhus Sygehus, Aarhus N, Jutland
  - Odense Universitetshospital, Odense C, Syd
- France (11):
  - Institut Bergonié - Centre Régional de Lutte Contre Le Cancer de Bordeaux et Sud Ouest, Bordeaux, Aquitaine
  - Hopital de la Pitie Salpetriere, Paris, Cedex 13
  - Hôpital Saint Vincent-de-Paul, Lille, Hauts-de-France
  - Chu De Nancy Hop D'Adultes De Brabois, Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - Pole Regionalde Cancérologie(CHU de Poitiers), Politiers, Politiers
  - Centre de Lutte Contre le Cancer - Centre Henri Becquerel Normandie Rouen, Rouen, Seine-Maritime
  - Centre Hospitalier Universitaire de Nantes - L' Hopital l'hôtel-Dieu, Nantes
  - Institut Curie, Paris
  - Centre hospitalier universitaire de Haut Leveque, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHRU De Tours, Tours
- Germany (8):
  - Universitätsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Klinikum der Universität München Großhadern, Würzburg, Bavaria
  - Universitätsklinikum Gießen und Marburg GmbH, Giessen, Hesse
  - Universitätsklinikum Münster - Albert Schweitzer Campus, Münster, North Rhine-Westphalia
  - InVO Institut für Versorgungsforschung in der Onkologie, Koblenz, Rhineland-Palatinate
  - Universitätsmedizin Johannes Gutenberg Universität Mainz, Mainz, Rhineland-Palatinate
  - Universitätsklinikum Schleswig-Holstein, Lübeck, Schleswig-Holstein
  - OncoResearch Lerchenfeld GmbH, Hamburg
- Israel (4):
  - Bnai Zion Medical Center, Haifa
  - Hadassah Medical Center, Jerusalem
  - Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (10):
  - Presidio Ospedaliero Civile Santi Antonio e Biagio, Alessandria, AL
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola, Emilia-Romagna
  - Ospedale Santa Maria delle Croci, Ravenna, Emilia-Romagna
  - Ospedale San Raffaele, Milan, Lombardy
  - IRCCS - AOU di Bologna, Bologna
  - IRCCS Ospedale Policlinico San Martino, Genova
  - Ospedale Vincenzo Cervello, Palermo
  - Irccs Crob, Potenza
  - Arcispedale Santa Maria Nuova, Reggio Emilia
  - Ospedale Di Circolo E Fondazione Macchi, Varese
- Japan (12):
  - Nagoya Medical Center, Nagoya, Aichi-ken
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Tohoku University Hospital, Sendai, Miyagi
  - Kindai University Hospital, Osaka Sayama-shi, Osaka
  - Saitama Medical Center, Kawagoe, Saitama
  - Japanese Foundation for Cancer Research, Koto, Tokyo
  - Chugoku Central Hospital, Hiroshima
  - Kumamoto University Hospital, Kumamoto
  - Kyoto Furitsu Medical University Hospital, Kyoto
  - Okayama University Hospital, Okayama
- Netherlands (3):
  - Bravis Ziekenhuis, Bergen op Zoom, North Brabant
  - Erasmus Medisch Centrum, Rotterdam
  - Ziekenhuisapotheek HagaZiekenhuis, The Hague
- New Zealand (2):
  - Christchurch Hospital, Addington, Christchurch
  - Middlemore Clinical Trials, Auckland
- Poland (6):
  - Centrum Onkologii Ziemi Lubelskiej, Lublin, Lublin Voivodeship
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Pratia MCM Krakow, Krakow
  - Wojewódzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii, Lodz
  - AIDPORT Sp. z o.o., Skorzewo
  - Uniwersytecki Szpital Kliniczny Klinika, Wroclaw
- Portugal (2):
  - IPOFG - Lisboa, Lisbon
  - Champalimaud Foundation, Lisbon
- Russia (3):
  - GUZ of Moscow City Clinical Hospital n.a. S.P. Botkin, Moscow
  - Fed. State Budgetary Institution "Russian Scientific & Research Institute of Hemat. & Transfusiology of Fed. Medico-Bio. Agency, Saint Petersburg
  - State Medical University named after I.P. Pavlov, Saint Petersburg
- South Korea (5):
  - Gachon University Gil Medical Center, Namdong-gu, Incheon-gwangyeoksi [Incheon]
  - Seoul National University Hospital, Seoul, Korea
  - Kosin University Gospel Hospital, Busan, Seogu
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul-teukbyeolsi [Seoul]
  - Asan Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
- Spain (11):
  - Hospital Universitario Virgen de la Victoria, Málaga, Andalusia
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [Barcelona]
  - Hospital Duran I Reynals, L'Hospitalet de Llobregat, Barcelona
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital Universitario Son Espases, Palma de Mallorca, Palma de Mallorca(Baleares)
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clínico Universitario de Valencia, Valencia
- Kantonsspital Luzern, Lucerne, Canton of Lucerne, Switzerland
- Taiwan (8):
  - Tri-Service General Hospital, Taipei City, Taipei
  - Chang Gung Memorial Hospital - Chiayi, Chiayi County
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng-Kung Uni. Hosp., Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital - Linkou, Taoyuan
- United Kingdom (7):
  - Aberdeen Royal Infirmary, Aberdeen, Aberdeen City
  - Derriford Hospital, Plymouth, Devon
  - GenesisCare, Newmarket, Suffolk
  - Beatson West of Scotland Cancer Centre, Glasgow
  - City Hospital, Nottingham University Hospitals, Nottingham
  - Churchill Hospital, Oxford
  - GenesisCare, Windsor, Windsor

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eyre TA, Shah NN, Dreyling M, Jurczak W, Wang Y, Cheah CY, Song Y, Gandhi M, Chay C, Sharman J, Andorsky DJ, Messersmith HM, Ruppert AS, Muthig VA, Ito R, Wang ML. BRUIN MCL-321: phase III study of pirtobrutinib versus investigator choice of BTK inhibitor in BTK inhibitor naive mantle cell lymphoma. Future Oncol. 2022 Nov;18(36):3961-3969. doi: 10.2217/fon-2022-0976. Epub 2022 Nov 15. PMID 36377973